CLINICAL TRIAL: NCT04562805
Title: Infinity-Swedeheart Study: Registry Based Randomized Clinical Trial (R-RCT) Comparing Long Term Outcomes of the DynamX Bioadaptor to the Resolute Onyx Stent in a More-comer PCI Patient Population
Brief Title: Infinity-Swedeheart Registry Based Randomized Clinical Trial (R-RCT)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Elixir Medical Corporation (Industry)
Collaborators: Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ELX-CL-1806
Record Dates: First submitted 2020-09-15; First posted 2020-09-24 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Coronary Artery Disease; Ischemic Heart Disease
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Ischemia

STUDY DESIGN:
Who Masked: Participant
Masking Description: The patients will be blinded to the assigned device from the point of randomization onward. Study site personnel will be trained not to disclose the treatment assignment to the patient. Site personnel assigned to conduct phone follow-up visits will be provided with a standard interview script in order to reduce bias.
  The Clinical Event Committee will be blinded to the fullest extent possible with only redacted source documents included in the event packages.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- DynamX Bioadaptor (Experimental): Elixir Medical DynamX™ Sirolimus Eluting Coronary Bioadaptor
  Interventions: Device: DynamX Bioadaptor
- Medtronic Resolute Onyx Stent (Active Comparator): Medtronic Resolute Onyx™ Zotarolimus-Eluting Coronary Stent System
  Interventions: Device: Resolute Onyx

INTERVENTIONS:
Device: DynamX Bioadaptor — DynamX Bioadaptor Treatment
  Arms: DynamX Bioadaptor
Device: Resolute Onyx — Resolute Onyx Treatment
  Arms: Medtronic Resolute Onyx Stent

SUMMARY:
The Infinity-Swedeheart trial is a prospective, multicenter, single-blind, randomized registry-based clinical trial. Eligible patients will be randomized 1:1 (DynamX Bioadaptor : Resolute Onyx).

DETAILED DESCRIPTION:
The Infinity-Swedeheart trial is a prospective, multicenter, single-blind, randomized registry-based clinical trial. Eligible patients will be randomized 1:1 (DynamX Bioadaptor : Resolute Onyx). 2400 Patients will be randomized in Sweden. Patients will be followed at 30 days and 1 year by phone, and at 6 months and 2 to 5 years through clinical and diagnostic registries.

ELIGIBILITY:
General Inclusion Criteria:

* Patient age ≥ 18 and ≤ 85 years
* Patient understands the trial requirements and treatment procedures and provides informed consent prior to any trial-specific tests or treatment
* Patients with CCS (stable angina, chronic angina, and chronic coronary artery disease) or ACS (unstable angina, ST-elevated myocardial infarction, and non-ST-elevated myocardial infarction) indicated for a percutaneous intervention with stent implantation.

Angiographic Inclusion Criteria:

* Patient has ≤ 3 lesions planned to be treated during the index procedure, each in a native epicardial vessel (including up to 1 planned Non-Target Lesion).

  1. Treatment is limited to a maximum of 2 Target Lesions per epicardial vessel. Any planned Non-Target Lesion must be located in a separate vessel from Target Lesion(s).
  2. When treatment of 2 target lesions in a single epicardial vessel is planned, there must be adequate separation between lesions to ensure a gap of greater than or equal to 10 mm between study devices.
  3. If a planned Non-Target Lesion is present it must have been treated without complication* prior to randomization.
  4. The definition of epicardial vessels is the LAD, LCx and RCA, and is inclusive of their branches.
* Target Lesion vessel diameter(s) and lesion length(s) suitable for implantation with either study device (DynamX Bioadaptor or Control) using a single device per lesion.
* Successful pre-dilatation of a minimum of 1 Target Lesion, defined as no waist in the inflated pre-dilatation balloon (using two orthogonal views) with a pre-dilatation balloon diameter size approximately 0.25 mm smaller than reference vessel diameter but not more than 0.5 mm smaller than the reference vessel diameter. A residual diameter stenosis prior to study device implantation by visual estimate is recommended to be < 30%.

General Exclusion Criteria:

* Acute myocardial infarction with Killip class III and IV
* Known history of chronic heart failure with LVEF < 30%
* Life expectancy < 2 years
* Patients on renal dialysis or with known eGFR < 30 ml/min
* Planned surgery necessitating interruption of dual antiplatelet therapy within 6 months after the index procedure
* Known intolerance to components of the study device or control stent or medication required (e.g. intolerance to concomitant anticoagulation or antiplatelet therapy)
* Patient has a current diagnosis of active COVID-19 disease
* Patient is currently participating in another clinical trial with an investigational device or an investigational drug that has the potential to impact study results (such as, anti-thrombotic or anti-platelet medications) that has not yet completed its primary endpoint
* Known pregnancy or breastfeeding
* Patient is, in the opinion of the Investigator, unable to comply with the requirements of the study protocol or is unsuitable for the study for any reason
* Subject has undergone prior PCI in a target vessel during the last 12 months. (A target lesion can be randomized and treated if a vessel contains a stent older than 12 months if the stent is more than 10 mm from the intended target lesion.)

Angiographic Exclusion Criteria:

* Lesions in the left main artery
* Venous or arterial bypass grafts
* In-stent restenosis
* Chronic total occlusion
* Ostial lesions (< 3 mm of the ostium of the RCA, LAD or LCx)
* Prior stent located in a Non-Target Vessel < 48 hours prior to the index procedure
* Lesion with severe calcification and/or tortuosity requiring the planned use of a guide extension catheter, rotablation or atherectomy
* Bifurcation lesions requiring a planned 2 or more stent technique

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2400 (Estimated)
Dates: Start 2020-09-30 (Actual); Primary Completion 2024-09-05 (Actual); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Target Lesion Failure (TLF) | 1 year
  Device Oriented Clinical Endpoint (DOCE) of target lesion failure (TLF; cardiovascular death, target vessel myocardial infarction (TV-MI), or ischemia-driven target lesion revascularization (ID-TLR))

SECONDARY OUTCOMES:
Landmark Analysis | 5 years or at the conclusion of the study
  DOCE from 6 Months to End of Follow-Up, DOCE of TVF from 6 Months to End of Follow-Up, DOCE from 6 Months to End of Follow-Up in subjects with ACS at Baseline
Device Success | During Study Procedure
  Lesion-Level Analysis
Procedural Success | In-Hospital, assessed up to 7 days
  Patient-Level Analysis
Composite Rate of Device Oriented Clinical Endpoint (DOCE) | 30 days, 6 months, 1-5 years
  Composite Device Oriented Clinical Endpoint (DOCE) (TLF; cardiovascular death, TV-MI, ischemia-driven TLR)
Composite Rate of Patient Oriented Clinical Endpoint (POCE) | 30 days, 6 months, 1-5 years
  Composite Patient Oriented Clinical Endpoint (POCE) (all-cause mortality, any stroke, any myocardial infarction (includes non-target vessel territory) and any revascularization). Note: Stroke to be collected and included in the POCE at 1 year and 5 years only.
Rate of Target Vessel Failure (TVF) | 30 days, 6 months, 1-5 years
  Target vessel failure (TVF; cardiovascular death, target vessel myocardial infarction (TV-MI), or target vessel revascularization (TVR))
Composite Rate of cardiovascular death, any myocardial infarction and any revascularization | 30 days, 6 months, 1-5 years
  Composite of cardiovascular death, any myocardial infarction and any revascularization
Rate of Ischemia driven target lesion revascularization (ID-TLR) | 30 days, 6 months, 1-5 years
  Ischemia driven target lesion revascularization (ID-TLR)
Rate of Target Lesion Revascularization (TLR) | 30 days, 6 months, 1-5 years
  All Target Lesion Revascularization
Rate of Target Vessel Revascularization (TVR) | 30 days, 6 months, 1-5 years
  All Target Vessel Revascularization
Rate of Ischemia driven target vessel revascularization (ID-TVR) | 30 days, 6 months, 1-5 years
  Ischemia driven target vessel revascularization (ID-TVR)
Rate of Ischemia driven non target vessel revascularization (ID-NTVR) | 30 days, 6 months, 1-5 years
  Ischemia driven non target vessel revascularization (ID-NTVR)
Rate of Non target vessel revascularization (NTVR) | 30 days, 6 months, 1-5 years
  Non target vessel revascularization (NTVR)
Rate of All revascularization | 30 days, 6 months, 1-5 years
  All revascularization
Rate of Myocardial Infarction | 30 days, 6 months, 1-5 years
  All MI, Q-Wave and Non Q-Wave MI, TV-MI, NTV-MI
Rate of Death | 30 days, 6 months, 1-5 years
  Cardiovascular Death, All-Cause Death
Composite: Cardiovascular death or myocardial infarction | 30 days, 6 months, 1-5 years
  Composite: Cardiovascular death or myocardial infarction
Composite: All-cause death or myocardial infarction | 30 days, 6 months, 1-5 years
  Composite: All-cause death or myocardial infarction
Composite: All-cause death, myocardial infarction or target vessel revascularization | 30 days, 6 months, 1-5 years
  Composite: All-cause death, myocardial infarction or target vessel revascularization
Rate of any stroke | 1 year and 5 years
  Any stroke (collected at 1 year and 5 years only)
Anginal Status | 30 days, 1,3,4 and 5 years
  Anginal Status by Seattle Angina Questionnaire-7 (SAQ-7)
Rate of Stent Thrombosis | 30 days, 6 months, 1-5 years
  Composite: Probable or definite stent thrombosis Probable Stent Thrombosis Definite Stent Thrombosis

CONTACTS AND LOCATIONS:
Overall Officials: David Erlinge, MD, PhD, Principal Investigator — Skane University Hospital, Lund; Stefan James, MD, PhD, Study Chair — Uppsala University
Locations (19):
- Sweden (19):
  - Mälarsjukhuset Eskilstuna, Eskilstuna
  - Hallands sjukhus, Halmstad
  - Helsingborgs lasarett, Helsingborg
  - Blekingesjukhuset i Karlskrona, Karlskrona
  - Centralsjukhuset Karlstad, Karlstad
  - Skånes Universitetssjukhus i Lund, Lund
  - Skånes Universitetssjukhus i Malmö, Malmo
  - Universitetssjukhuset Örebro, Örebro
  - Östersunds sjukhus, Östersund
  - Sunderby sjukhus, Södra Sunderbyn
  - Capio St Görans sjukhus, Stockholm
  - Danderyds sjukhus, Stockholm
  - Karolinska Universitetssjukhuset Huddinge, Stockholm
  - Karolinska Universitetssjukhuset Solna, Stockholm
  - Södersjukhuset, Stockholm
  - Sundsvall Hospital, Sundsvall
  - Norrlands universitetssjukhus Umeå, Umeå
  - Akademiska Sjukhuset, Uppsala
  - Västmanlands sjukhus i Västerås, Västerås

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Erlinge D, Andersson J, Frobert O, Tornerud M, Hamid M, Kellerth T, Grimfjard P, Winnberg O, Jurga J, Wagner H, Zwackman S, Adielsson M, Alstrom P, Masoe E, Ulvenstam A, Millgard J, Bohm F, Held C, Renlund H, Oldgren J, Smits PC, Elek C, Abizaid A, James S. Bioadaptor implant versus contemporary drug-eluting stent in percutaneous coronary interventions in Sweden (INFINITY-SWEDEHEART): a single-blind, non-inferiority, registry-based, randomised controlled trial. Lancet. 2024 Nov 2;404(10464):1750-1759. doi: 10.1016/S0140-6736(24)02227-X. Epub 2024 Oct 28. PMID 39481425